CLINICAL TRIAL: NCT05110352
Title: Pilot Epidemiological Study to Determine the Prevalence of Pharyngolaryngeal Reflux in Patients Treated for Obstructive Sleep Apnea Syndrome
Brief Title: Prevalence of Pharyngolaryngeal Reflux in Patients Treated for Obstructive Sleep Apnea Syndrome
Acronym: RESTECH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A02789-30
Record Dates: First submitted 2021-10-21; First posted 2021-11-05 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Obstructive Sleep Apnea; Reflux, Laryngopharyngeal
MeSH Terms: conditions — Sleep Apnea, Obstructive; Laryngopharyngeal Reflux | interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obstructive Sleep Apnea Syndrome patients with polysomnography planned (Experimental): Apnea-Hypopnea Index (AHI) > 15
  Interventions: Diagnostic Test: Polysomnography; Diagnostic Test: Pharyngeal ph-metry Restech; Procedure: Peptest; Behavioral: Questionnaire RSS-12; Procedure: Reflux Sign Assessment

INTERVENTIONS:
Diagnostic Test: Polysomnography — A polysmnography is planned for every patients in order to evaluate the Apnea-Hypopnea Index (AHI).
Diagnostic Test: Pharyngeal ph-metry Restech — Pharyngeal ph-metry Restech over 24 hours (night and day)
Procedure: Peptest — Saliva sample to look for an association between pharyngolaryngeal reflux and obstructive sleep apnea syndrome
Behavioral: Questionnaire RSS-12 — Questionnaire with 12 items about quality of life. Score between 0 and 5.
Procedure: Reflux Sign Assessment — RSA score about anatomy and morphology of the mouth

SUMMARY:
The aim of the study is to find, using validated and efficient tools, a laryngopharyngeal reflux in patients receiving polysomnography for suspected obstructive sleep apnea syndrome.

It is proposed to carry out simultaneously, at the Sleep Center of the Polyclinique of Poitiers (CSPP), a polysomnography, a 24-hour Restech pharyngeal pH-metry (day and night), a Peptest (in the evening and in the morning of the polysomnography), with the RSS-12 questionnaire and the RSA score.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 ans)
* Polysomnography planned for OSA assessment
* RPL known or not, suspected or not
* Affiliation to a social security scheme or beneficiary of such a scheme
* Patient having signed the free and informed consent

Exclusion Criteria:

* Minors
* Smoking, alcoholism, chronic or serious disabling pathology
* Medical history of upper aerodigestive tract cancer, radiotherapy
* Recent infection of upper aerodigestive tract, chronic rhinosinusitis
* Permanent nasal obstruction
* Active allergy
* Non-obstructive SAS (central)
* Patient under anti-secretory treatment (IPP) during the 8 days preceding the Restech associated with the PSG
* Refusal to participate in the study
* Protected patients: Adults under guardianship, guardianship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, breastfeeding or parturient
* Hospitalized without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-04-23 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Obstructive Sleep Apnea Syndrome diagnosed with pharyngolaryngeal reflux. | 3 months
  the diagnosis of OSA is posed by the PSG as soon as the AHI is ≥ 15 / h

SECONDARY OUTCOMES:
RSS-12 score | 3 months
  Positive (>11)
RSA score | 3 months
  Positive if > 14
Peptest | 3 months
  Positive if > 75 ng / mL

CONTACTS AND LOCATIONS:
Locations (1):
- Centre du Sommeil de la Polyclinique de Poitiers, Potiers, France